CLINICAL TRIAL: NCT05134077
Title: Influence of Simple Renal Cysts on Renal Function: Cohort Clinical Trial.
Brief Title: Influence of Simple Renal Cysts on Renal Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Moscow State University of Medicine and Dentistry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SRC
Record Dates: First submitted 2021-10-19; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Simple Renal Cyst; Renal Function Disorder
Keywords: Simple Renal Cyst, Renal Function
MeSH Terms: interventions — Contrast Media

STUDY DESIGN:
Intervention Model Description: We present a cohort study of patients with renal cysts (the first group - kidneys with cysts, the second group - kidneys without cysts in the studied patients). All patients will undergo contrast-enhanced CT of the urinary system (volume of atrophic parenchyma will be calculated), as well as nephroscintigraphy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kidneys with simple cysts (Experimental): Patients involve from Citi Clinical Hospital with simple renal accidentally discovered cyst.
  Interventions: Procedure: CT scan with contrast; Radiation: Nephroscintigraphy
- contralateral kidneys without cyst (Active Comparator): Рatients involve from Citi Clinical Hospital with simple renal accidentally discovered cyst.
  Interventions: Procedure: CT scan with contrast; Radiation: Nephroscintigraphy

INTERVENTIONS:
Procedure: CT scan with contrast — CT scan with contrast is necessary to determine the position of renal cysts, their location, and size (determine volume of atrophic parenchyma will be calculated).
Radiation: Nephroscintigraphy — Nephroscintigraphy is necessary to determine the renal function

SUMMARY:
This is a prospective, cohort, randomized clinical trial examining the effect of simple renal cysts on renal function.

DETAILED DESCRIPTION:
This study is planned to include patients from S.I. Spasokukotskiy Citi Clinical Hospital with simple renal accidentally discovered cyst.

The aim of the study is to evaluate the impact of simple renal cysts on renal function and explore the correlation between cyst's size, parenchymal atrophy, and renal function.

After receiving the results, the analysis of the data obtained is carried out.

1. The symmetry of the function of both kidneys is analyzed
2. The relationship between the presence of a simple kidney cyst and a decrease in its function in comparison with a healthy kidney is analyzed.
3. The relationship between the maximum size of a kidney cyst and a decrease in its function in comparison with a healthy kidney is analyzed.
4. The relationship between the volume of the atrophied kidney parenchyma and a decrease in its function as compared with a healthy kidney is analyzed.
5. Correspondence of GFR indices obtained by scintigraphy and by calculation using the Schwartz formula

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with simple kidney cyst Bosniak 1-2
* Normal blood creatinine values

Exclusion Criteria:

* Impossibility of performing CT with intravenous contrast enhancement.
* Bosniak 3-4
* CKD
* Bilateral cysts
* Multiple renal cysts
* Sinus cysts
* Cysts with a max size less than 2 cm.
* Single kidney
* Chronic kidney disease and conditions associated with the potential decrease of kidney function
* Glomerulonephritis
* Chronic pyelonephritis
* Amyloidosis
* Diabetes
* Autoimmune diseases
* Urolithiasis
* Kidney and upper urinary tract surgery
* Anomalies of the kidneys and upper urinary tract with impaired outflow
* Calcification of the renal arteries
* Renal artery stenosis
* Hypertensive nephropathy
* Severe concomitant diseases requiring
* Chemotherapy
* Long-term (more than 10 days) antibiotic therapy in the last month
* Long-term (more than 7 days) use of NSAIDs in the last month
* Diagnostic and therapeutic manipulations accompanied by the introduction of X-ray contrast agents
* Secondarily shriveled or non-functioning kidney
* Kidney hypoplasia
* Accessory kidney
* a decrease in GFR below normal values for a kidney without a cyst (as determined by nephroscintigraphy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-02-16 (Estimated); Primary Completion 2022-03-08 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Renal function | 1 month
  Glomerular filtration rate (GFR, ml/min/1.73 m2) is a test used to check how well the kidneys are working. Specifically, it estimates how much blood passes through the glomeruli each minute. A GFR of 60 or higher is in the normal range. A GFR below 60 may mean kidney disease. A GFR of 15 or lower may mean kidney failure.
  The measurement of the glomerular filtration rate will be measured according to the results of the blood test and the results of nephroscintigraphy

SECONDARY OUTCOMES:
Ratio of cyst size and volume of atrophic renal parenchyma | 1 month
  Computed tomography with contrast will be used to determine the position of renal cysts, their location, size and volume of atrophic parenchyma (cm2) are calculated

CONTACTS AND LOCATIONS:
Overall Officials: Tukhtasin Mahmudov, Principal Investigator — Moscow state university of medicine and dentistry named after A.I. Evdokimov